CLINICAL TRIAL: NCT02895035
Title: Prospective Comparison of Epinephrine and Phenylephrine/Ketorolac (Omidria®) Additives With Regards to Intraoperative Pupil Size
Brief Title: Comparison of Epinephrine and Phenylephrine/Ketorolac With Regards to Pupil Size
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Data analysis was never performed by sub-investigator
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Seth M Pantanelli, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 00005630
Record Dates: First submitted 2016-09-04; First posted 2016-09-09 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epinephrine (Active Comparator): Epinephrine is the intracameral additive during cataract surgery.
  Interventions: Drug: Epinephrine
- Omidria (Active Comparator): Omidria is the intracameral additive during cataract surgery.
  Interventions: Drug: Phenylephrine-ketorolac

INTERVENTIONS:
Drug: Phenylephrine-ketorolac — Pehnylephrine-ketorolac is a combination of an alpha-one agonist (phenylephrine) and an NSAID (ketorolac). One 4-mL bottle of 1% phenylephrine/3% ketorolac is added to the irrigation solution during cataract surgery.
  Other Names: Omidria
  Arms: Omidria
Drug: Epinephrine — Epinephrine is a nonselective adrenergic agonist added to the irrigation solution during cataract surgery.
  Arms: Epinephrine

SUMMARY:
The objective of this study is to compare the maintenance of intraoperative mydriasis during cataract surgery between two drugs: epinephrine, which has routinely been used for decades, and Omidria, a newly FDA approved combination drug of phenylephrine and ketorolac. Patients undergoing cataract surgery that are enrolled in the trial will randomly receive one of the drugs in one eye, and the other eye will receive the drug during the subsequent cataract surgery.

DETAILED DESCRIPTION:
Cataract remains a leading cause of correctable blindness worldwide. Over 3.5 million cataract surgeries in the United States and 20 million cataract surgeries worldwide are performed every year. Cataract surgery is performed by making a small incision, removing the cataractous lens, most often through the process of phacoemulsification, and replacement with an intraocular lens. Like all surgeries, adequate exposure and field of view is vital for a safe and effective surgery. In cataract surgery, the field of view is limited by the diameter of the pupil. Several different drugs, such as cyclopentolate, tropicamide, phenylephrine, and epinephrine are utilized to maintain dilation (mydriasis) of the pupil during surgery.

There are currently two prospective randomized controlled trials comparing phenylephrine/ketorolac to placebo in the published literature. Both of these studies demonstrated that phenylephrine/ketorolac is superior to placebo for the maintenance of mydriasis during cataract surgery. Epinephrine has been the standard of care for intraoperative mydriasis. Phenylephrine/ketorolac (Omidria) is a newly FDA-approved additive for the maintenance of intraoperative mydriasis, but there are currently no published studies comparing epinephrine to phenylephrine/ketorolac for maintenance of mydriasis during cataract surgery.

While both of these drugs have been shown to be superior to placebo for the maintenance of mydriasis, there is a significant cost difference between epinephrine, which has been used for many years, and phenylephrine/ketorolac, which gained FDA approval in 2014. One 4 mL vial of Omidria® is utilized for one cataract surgery, which costs $465.

The primary endpoint to be measured in the study is the mean area under the curve change from baseline in pupil diameter over time to the end of cataract surgery.

Secondary endpoints will be maximum intraoperative pupil constriction, subjects with pupil diameter less than 6.5 mm at any during surgery, subjects with pupil less than 6.0 mm during cortical clean-up, and subjects with greater than 2.5 mm of pupillary constriction at any time during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are older than 18 years of age
* Patients who are planned to undergo bilateral cataract surgery
* Patients with baseline IOP of 5 - 22 mm Hg
* Medicare insurance*

  * There is a significant cost difference between our two study drugs. Therefore, Medicare insurance is part of our inclusion criteria, because there is a pass-through reimbursement in place to cover the cost of phenylephrine/ketorolac. Other insurances (for example, Aetna Better Health, Highmark Freedom, Gateway) have variable or poor coverage for phenylephrine/ketorolac, which would leave the medical center responsible for the cost. Patients can never be held responsible for the cost of the medication because it is included in "covered services" for cataract surgery billing.

Exclusion Criteria:

* Patients who are planned to undergo only unilateral cataract surgery
* Patients who are planned to undergo cataract surgery and another surgical procedure in the same operation (eg. combined cataract and glaucoma surgery)
* Patients with concurrent clinically significant disease, connective tissue disease, abnormal blood pressure at screening, narrow-angle or unstable glaucoma or treatment with prostaglandins, uncontrolled chronic eye disease or active corneal pathology or scarring
* Patients with history of iritis or trauma with iris damage
* Patients with recent eye surgery (non-laser surgery within 3 months or laser surgery within 30 days prior to study surgery)
* Patients with clinically significant hypersensitivity to the study medications
* Patients who have used pilocarpine (a pupil constrictor) within 6 months prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients who presented to one of two attending ophthalmologist's (MCC or SMP) clinics at Penn State Eye Center for cataract evaluation between November 10, 2016 and February 8, 2018 and met inclusion/exclusion criteria were invited to participate in the study. There were no incentives provided to patients for enrolling in the study.
Groups:
- Epinephrine (1 Day), Washout (21 Days), Then Omidria (1 Day): Patients in this arm received epinephrine during the first eye surgery. Patients then waited (washout) 21 days before proceeding with second eye surgery. Patients then received Omidria during the second eye surgery.
- Omidria (1 Day), Washout (21 Days), Then Epinephrine (1 Day): Patients in this arm received Omidria during the first eye surgery. Patients then waited (washout) 21 days before proceeding with second eye surgery. Patients then received epinephrine during the second eye surgery.
Period: Overall Study
Arm/Group | Epinephrine (1 Day), Washout (21 Days), Then Omidria (1 Day) | Omidria (1 Day), Washout (21 Days), Then Epinephrine (1 Day)
Started | 23 | 36
Completed | 18 | 24
Not Completed | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All Participants were randomized to receive all interventions. Therefore, the baseline characteristics are grouped as "all participants"
Arm/Group | All Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42
Tamsulosin Use [Count of Participants; unit: Participants]
  Tamsulosin | 1
  No Tamsulosin | 41

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve Change From Baseline in Pupil Diameter Over Time to the End of Cataract Surgery
Description: Mean area under the curve was calculated by assessing the pupil diameter at baseline and then again at 1 minute intervals until the surgery was complete (max 20 minutes). Units are in millimeters*seconds
Time Frame: During cataract surgery, with maximum end time of 20 minutes
Population: Two eyes from each participant were included for all outcome measures.
Measure: Mean (Standard Deviation); unit: millimeters * seconds
Units Other Than Participants: Eyes
Arm/Group | Epinephrine | Omidria
Number analyzed (Participants) | 42 | 42
Number analyzed (Eyes) | 42 | 42
millimeters * seconds | 1.76 (6.51) | 0.8 (12.01)

2. Secondary Outcome: Maximum Intraoperative Change in Pupil Diameter
Description: This is the maximum observed change in pupil diameter, as measured compared to baseline.
Time Frame: During cataract surgery, with maximum end time of 20 minutes
Population: Two eyes from each participant were included
Measure: Mean (Standard Deviation); unit: millimeters
Units Other Than Participants: Eyes
Arm/Group | Epinephrine | Omidria
Number analyzed (Participants) | 42 | 42
Number analyzed (Eyes) | 42 | 42
millimeters | -0.71 (0.57) | -0.66 (0.79)

3. Secondary Outcome: Number of Eyes With Pupil Diameter Less Than 6 mm at Any Time During Surgery
Description: Number of eyes with a measured pupil diameter less than 6 mm at any time during surgery
Time Frame: During cataract surgery, with maximum end time of 20 minutes
Population: Each participant had two eyes included in the study
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Epinephrine | Omidria
Number analyzed (Participants) | 42 | 42
Number analyzed (Eyes) | 42 | 42
Eyes | 3 | 2

4. Secondary Outcome: Number of Eyes With Pupil Diameter Less Than 6 mm During Cortical Clean-up
Description: Number of eyes with a measured pupil diameter less than 6 mm during cortical clean-up
Time Frame: During cataract surgery, cortical clean-up stage, up to 5 mins
Population: Each participant had two eyes included in the study
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Epinephrine | Omidria
Number analyzed (Participants) | 42 | 42
Number analyzed (Eyes) | 42 | 42
Eyes | 3 | 2

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Epinephrine | Omidria
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
small sample size some patients received pre-operative topical NSAID in both eyes, while others did not

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT02895035/Prot_SAP_000.pdf